CLINICAL TRIAL: NCT00473018
Title: Behavioral, Clinical and Basic Science Studies of Non-occupational Post-exposure Prophylaxis ("PEP-2")
Acronym: PEP-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 5R01MH061180 (NIH)
Record Dates: First submitted 2007-05-09; First posted 2007-05-14 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2007-05

CONDITIONS: HIV Infections
Keywords: postexposure prophylaxis; HIV Seronegativity
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: standard versus enhanced risk reduction counseling

SUMMARY:
This is a randomized trial to compare the effect of standard versus enhanced risk reduction counseling on risk behavior incidence in individuals receiving PEP medications. The study seeks to 1) determine if there are equivalent changes in the incidence of self-reported risk behaviors, STD incidence, and adherence to medications in individuals who receive enhanced risk reduction and adherence counseling and those who received standard risk reduction and adherence counseling; 2) evaluate viral and host biological factors involved in sexual transmission that may either influence PEP efficacy, or themselves be negatively or positively affected by the administration of PEP medications; and 3) contribute to the CDC registry in an attempt to provide crucial data for a case control analysis to establish the efficacy of PEP for sexual and injection drug use exposures. The principal outcome will be the change in participants' number of unprotected sexual acts following administration of PEP. This is defined as the number of prior 3-month acts of high risk unprotected sex, assessed at 12 months following a course of PEP, minus the number of unprotected acts the participant reported in the 3 and 6 months prior to beginning PEP (assessed at baseline). Methods to be used consist of interview data collection, questionnaires, risk reduction and adherence counseling and source recruitment counseling (index subject).

DETAILED DESCRIPTION:
A. SPECIFIC AIMS Our group (including behavioral, epidemiological, basic, and clinical scientists from UCSF, San Francisco General Hospital, The San Francisco Department of Public Health, and the UCSF-affiliated Gladstone Institute of Virology and Immunology) conducted a feasibility study of Post Exposure Prevention (PEP) in which we successfully recruited, retained, and assessed over 400 individuals recently and substantially exposed to HIV-1 (index cases), as well as a significant number of the persons (source cases) who exposed the index cases to HIV-1.

We are frequently asked by physicians and public health professionals for help in establishing similar programs in various communities. PEP has two promising possibilities: (a) it may prevent HIV infection and (b) it may be a viable way to attract high risk uninfected individuals into counseling. But tremendous uncertainty remains about how to integrate PEP into existing clinical and prevention programs. Because we felt that risk reduction counseling was essential to prevent disinhibition, we provided intensive (5 session) prevention counseling in our feasibility study. Adherence counseling was also essential as incomplete adherence could reduce the effectiveness of the medications or increase the chance of infection with a resistant isolate. However, multi-session counseling is very resource intensive.

The most urgent question to be addressed about PEP is whether PEP medications must be offered with an enhanced counseling program, or if standard HIV pre- and post-test counseling and routine adherence counseling will result in equivalent risk behavior following PEP and adherence with antiretroviral medications.

Thus, we propose the following primary aim:

1. To conduct a randomized trial to determine whether enhanced (multi-session) risk reduction and adherence counseling is equivalent to standard (2 session) risk reduction and adherence counseling in terms of self-reported risk behaviors and documented STDs and adherence to PEP medications.

   In addition, because we are recruiting a cohort of HIV-infected individuals who are engaging in behavior potentially capable of transmitting HIV, as well as HIV uninfected individuals who have recently exposed themselves to HIV, we have the unique opportunity to address the following important aims:
2. Source (HIV infected person potentially transmitting) virologic characteristics: To describe and compare the (a) HIV-1 RNA level and (b) antiretroviral resistance mutation prevalence in the plasma and genital secretions of source subjects.
3. Index (exposed HIV uninfected) subject CD8+ T-cell antiviral factor activity responses:

   1. To determine whether PEP medications blunt CD8+ T-cell antiviral factor (CAF) activity by comparing the changes in CAF following HIV exposure in persons receiving PEP medications to individuals matched for exposure who do not receive medications;
   2. To determine whether there is a correlation between source plasma and genital secretion HIV-1 RNA levels and index CAF activity.)
4. To evaluate the safety of adding 2 doses of nevirapine to the existing medication regimens that are based on two nucleoside analogue reverse transcriptase inhibitors ¬+ a protease inhibitor.

ELIGIBILITY:
Inclusion Criteria:

To be included in the study the subject must be:

* >/= 14 years of age
* Able to give informed consent
* English- or Spanish-speaking
* Able to report risk of HIV exposure during the previous 72 hours defined as:

  * unprotected sex defined as:

    * unprotected receptive or insertive anal or vaginal sex without a condom (with or without ejaculation); or
    * protected receptive or insertive anal or vaginal intercourse with a condom which breaks or falls off during intercourse (with or without ejaculation); or
    * sharing of potentially contaminated injection drug use equipment; or
    * unprotected receptive oral sex with ejaculation; and this exposure was with a
  * high risk partner defined as:

    * known to be HIV-infected; or
    * is a man who has sex with men; or
    * is or has been an injection drug user; or
    * is a sex worker, or
    * the partner is anonymous, or
    * the partner is known to the subject but their sexual or injection drug use history is unknown.
  * Additional exposures will be considered if they involve potentially HIV-infected body fluids in contact with a mucous membrane or non-intact skin, at the discretion of the study clinician. The subject must report that he/she has never received antiretroviral medications for the treatment of established HIV infection nor been diagnosed with HIV infection. The subject must elect to initiate PEP medications.
* Index subjects will be allowed to enroll in the study up to four times in one year (re-PEP). They will be encouraged to participate in referrals for enhanced prevention services at the direction of the counseling supervisor. Subjects who enroll more than once will be given 2 additional counseling sessions for each re-enrollment episode designed to address issues related to on-going exposure.
* All women will be tested for pregnancy; if pregnant, they will still be offered enrollment in the study, with additional counseling provided by the Bay Area Perinatal Aids Center (BAPAC) at San Francisco General Hospital.

Exclusion Criteria:

Subjects will be excluded if they are:

* Unable to give informed consent
* Known to be infected with HIV by their report
* Unable to commit to or make follow-up visits.

Cases of sexual assault will be referred to rape counseling services. PEP may be offered as a non-study service in collaboration with the rape counseling services.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Michelle E Roland, Principal Investigator — University of California, San Francisco